CLINICAL TRIAL: NCT06722300
Title: Clinical Study on the Impact of Eradication of Oral Porphyromonas Gingivalis on the Prognosis of Early Esophageal Cancer After ESD Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Henan University of Science and Technology (Other)
Collaborators: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PGESCC002
Record Dates: First submitted 2024-08-23; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-04

CONDITIONS: Esophageal Cancer
Keywords: Esophageal Cancer；; ESD; Porphyromonas gingivalis
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- No.1 (No Intervention): Pg negative
- No.2 (Experimental): Patients with Pg infection
  Interventions: Device: Ultrasonic teeth cleaning plus Tinidazole microneedle patches applying
- No.3 (No Intervention)

INTERVENTIONS:
Device: Ultrasonic teeth cleaning plus Tinidazole microneedle patches applying — After gargling with compound chlorhexidine rinse or 3% hydrogen peroxide rinse for 1 minute, ultrasonic teeth cleaning was performed. After teeth cleaning, the wound was rinsed with 3% hydrogen peroxide and bleeding was stopped. After ultrasonic teeth cleaning, two metronidazole oral composite microneedle patches were immediately applied to the upper and lower gums near the inner side of the first molar, especially where the teeth were lost or damaged. The mouth was kept closed for 15 minutes. After the microneedles were fully degraded, the patient could leave the clinic.
  Arms: No.2

SUMMARY:
Porphyromonas gingivalis (Pg) is a representative pathogenic bacterium of periodontitis and is a Gram-negative anaerobic bacterium. Epidemiological studies suggest that periodontitis is positively correlated with the risk of gastrointestinal tumors such as esophageal cancer. Pg has been extensively studied due to its unique ability to invade epithelial cells and survive in host blood and tissues, and has been confirmed to be associated with esophageal cancer, pancreatic cancer, and oral cancer. Pg is enriched in esophageal cancer tissues and atypical hyperplasia lesions of esophageal mucosa, and is rarely found in corresponding non-tumor parts, cardiac cardia, and stomach. Treating normal esophageal mucosal epithelial cells with Pg medium can induce atypical hyperplasia. Chen et al found that the Pg infection rate in esophageal squamous cell carcinoma is as high as 57%. Gao S et al. used 16S rDNA PCR technology to detect 100 ESCC patients. The detection rate of Pg pan-antigen was 61% in tumor tissues, 12% in para-cancerous tissues, and was not detected in normal mucosal tissues. Studies have shown that Pg and Pg/Prevotella ratio in saliva can be used as reference indicators for the diagnosis of esophageal cancer. The abundance of Pg in saliva and dental plaque is associated with the development of esophageal squamous cell carcinoma and poor prognosis. High levels of Pg-specific antibodies in serum are an independent predictor of poor prognosis in esophageal squamous cell carcinoma. Gao et al.'s study found that Pg infection is closely related to local recurrence after endoscopic resection. Studies based on ESCC patients data, animal models and esophageal squamous cell carcinoma cell lines have confirmed that Pg promotes the occurrence and development of esophageal cancer, leads to resistance to neoadjuvant chemotherapy, and weakens the efficacy of anti-tumor treatment. In summary, whether the recurrence of early esophageal cancer after ESD can be controlled by removing Pg deserves further exploration.

To this end, based on the combined treatment of mechanical removal and antibacterial drugs, this study designed a method that combines ultrasonic tooth cleaning with tinidazole oral composite microneedle patches to completely remove oral Pg and evaluate the impact on the prognosis of early ESCC after ESD therapy by extra removal of oral Porphyromonas gingivalis.

DETAILED DESCRIPTION:
The new oral microneedle patch was developed by the Oncology Molecular Biology Laboratory of the First Affiliated Hospital of Henan University of Science and Technology. The patch consists of a dissolvable basement membrane part and a needle tip loaded with drugs and polylactic acid-co-glycolic acid microspheres. The base film of the new oral microneedle patch is made of 10% gelatin. 10% gelatin can solidify at room temperature and dissolve in a few minutes at body temperature. Antibiotics can be loaded directly into the gelatin-based membrane and released rapidly. The tip part is made of gelatin methacryloyl (GelMA) cross-linked by UV light. GelMA forms a hydrogel structure that gradually degrades and can be used as a carrier for sustained drug release. After applying the oral microneedle patch, the basement membrane quickly dissolves and releases the tinide file, which can effectively reduce the content of harmful bacteria in the oral cavity. The needle tip structure composed of GelMA can penetrate and stay in the gingival tissue, continuously releasing tinide files and cytokines to promote the repair of gingival tissue.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed esophageal cancer;
* Newly diagnosed patients who meet the absolute and relative indications for ESD;
* ECOG: 0～1;
* Expected survival ≥12 weeks;
* Receive ESD treatment within 28 days and meet R0 standards;
* The main organ functions are normal, that is, the following standards are met:

  1. Routine blood examination:

     a.HB≥90g/L; b.ANC≥1.5×10^9/L; c.PLT ≥80×10^9/L;
  2. Biochemical examination:

     1. ALB≥30g/L; b.ALT and AST≤2.5ULN; if there is liver metastasis, ALT and AST≤5ULN; c.TBIL≤1.5ULN;
* Women of childbearing potential must agree to use contraceptive measures (such as intrauterine devices, birth control pills or condoms) during the study and within 6 months after the end of the study; have a negative serum or urine pregnancy test within 7 days before study enrollment , and must be non-lactating patients; males should agree that they must use contraceptive measures during the study period and within 6 months after the end of the study period;
* The subjects voluntarily joined this study, signed the informed consent form, had good compliance, and cooperated with the follow-up.

Exclusion Criteria:

* Does not meet the above selection criteria;
* Patients with distant visceral metastasis;
* Pathological confirmation after ESD does not meet Tis, T1a, R0 or the depth of the lesion exceeds pSM1, and the depth of submucosal invasion is >200 μm;
* The lesions are ulcerated and poorly differentiated (poorly differentiated, undifferentiated);
* There is lymphovascular infiltration;
* Those who are allergic to tinidazole or have metabolic disorders;
* Patients who require warfarin anticoagulation and those who cannot quit drinking;
* Patients who cannot tolerate ultrasonic tooth cleaning;
* Pregnant or lactating women;
* Patients with other malignant tumors within 5 years (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix);
* Those who have a history of psychotropic drug abuse and are unable to quit or patients with mental disorders;
* Patients who have participated in other drug clinical trials within four weeks;
* Patients who, according to the researcher's judgment, have concomitant diseases that seriously endanger patient safety or affect the patient's completion of the study;
* Patients with recurrent oral ulcers or other oral diseases that affect oral flora;
* Patients with chronic infectious diseases or autoimmune diseases who require long-term or repeated application of antibacterial drugs or glucocorticoids; those deemed not suitable for inclusion by the researcher.
* The researcher believes that the applicant is not suitable for inclusion.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 856 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
recurrence-free survival (RFS) | up to 5 years
  From enrollment to the end of follow-up or the date of first documented progression

SECONDARY OUTCOMES:
overall survival (OS) | up to 5 years
  From randomization to the end of follow-up or the time of the death event
the safety of the intervention methods | up to 5 years
  From enrollment to the end of follow-up or the date of confirmed adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Shegan Gao, MD，pHD, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology
Locations (1):
- The Clinical Medical College, The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided
The researchers will decide whether to share based on the research data.